CLINICAL TRIAL: NCT00717158
Title: Evaluating Healthcare Utilization, Costs and Health-Related Outcomes of a Medical Nutrition Therapy Intervention on Obese Patients With Type 2 Diabetes - A Pilot Study
Brief Title: Lifestyle Intervention's Impact on Health Care Costs
Acronym: ICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Anne Wolf, Principal Investigator, University of Virginia School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8742; Am Dietetic Assoc 9336
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Health Behavior; Lifestyle; health care costs; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Health Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (No Intervention): Usual medical care. They received written healthy lifestyle information
  Interventions: Behavioral: Usual medical care
- 2 (Active Comparator): Intervention participants were assigned to one registered dietitian who they met with over a one year period for 6 session (four hours) of individual care, 6- one-hour group classes, and had monthly email contact for follow up and checking in
  Interventions: Behavioral: Lifestyle Case management

INTERVENTIONS:
Behavioral: Usual medical care
  Arms: I
Behavioral: Lifestyle Case management — Intervention participants were assigned to one registered dietitian who they met with over a one year period for 6 session (four hours) of individual care, 6- one-hour group classes, and had monthly email contact for follow up and checking in
  Arms: 2

SUMMARY:
The ICAN Pilot project aims to evaluate the differences in economic, clinical and quality of life outcomes of a nutrition intervention involving lifestyle case management and medical nutrition therapy by a registered dietitian compared to usual medical care in obese persons with type 2 diabetes. The intervention is aimed at moderate weight loss (> 5-10%), improvement in diet quality and an increase in physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2, calculated from measured weight and height.
* Type 2 diabetics on medication for their diabetes.
* Age 20 -60 years of age.
* Have phone.
* Fluency in reading, writing and comprehension of English
* Have Qualchoice as their primary health insurer.

Exclusion Criteria:

* Depression, BDI score > 20
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2001-05; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Health Care utilization and costs using claims data | one year

SECONDARY OUTCOMES:
Weight change | one year
Change in hemoglobin A1c | One Year
Work days lost | One year
Disability Days | One year
Change in quality of life | one year

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Wolf, MS, RD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- University of Virginia School of Medicine, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Wolf AM, Conaway MR, Crowther JQ, Hazen KY, L Nadler J, Oneida B, Bovbjerg VE; Improving Control with Activity and Nutrition (ICAN) Study. Translating lifestyle intervention to practice in obese patients with type 2 diabetes: Improving Control with Activity and Nutrition (ICAN) study. Diabetes Care. 2004 Jul;27(7):1570-6. doi: 10.2337/diacare.27.7.1570. PMID 15220230
- [Result] Wolf AM, Siadaty M, Yaeger B, Conaway MR, Crowther JQ, Nadler JL, Bovbjerg VE. Effects of lifestyle intervention on health care costs: Improving Control with Activity and Nutrition (ICAN). J Am Diet Assoc. 2007 Aug;107(8):1365-73. doi: 10.1016/j.jada.2007.05.015. PMID 17659904